CLINICAL TRIAL: NCT00582465
Title: Bone Mineral Density of Children and Adolescents With Systemic Lupus Erythematosus
Brief Title: Study to Evaluate the Natural History of Osteoporosis in Children and Adolescents With Systemic Lupus Erythematosus
Acronym: BMD
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H8994-14731
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Lupus

SUMMARY:
This is a study to determine if people with Lupus have weak bones.

Test which is a better method for detecting bone changes:

* Dual energy X-ray absorptiometry (DXA)
* Single energy quantitative computed tomography (SEQCT)

Evaluate whether weak bones are associated with things like medications or amount of fat and muscle.

DETAILED DESCRIPTION:
This is a longitudinal cohort study to evaluate the natural history of osteoporosis in children and adolescents with Systemic Lupus Erythematosus.

The specific Aims are:

* To compare the BMD of children and adolescents with Systemic Lupus Erythematosus to healthy controls utilizing Dual energy X-ray absorptiometry (DXA) and Single energy quantitative computed tomography (SEQCT). The following questions will be addressed at baseline:

What is the variation of BMD seen among subjects with Systemic Lupus Erythematosus? Is the BMD of children with Systemic Lupus Erythematosus diminished relative to healthy controls? If BMD is diminished, what is the severity of the reduction?

* To characterize the annual change in BMD for children and adolescents with Systemic Lupus Erythematosus over a five year period in a longitudinal cohort study utilizing arial and volumetric densitometry methods of both trabecular- and cortical-rich regions of bone.
* To compare the use of DXA and SEQCT for measuring BMD in children and adolescents with Systemic Lupus Erythematosus.
* To characterize the determinants of BMD and corresponding markers of bone metabolism in a longitudinal cohort of pediatric Systemic Lupus Erythematosus subjects.
* To bank Systemic Lupus Erythematosus subject blood and urine specimens for future analysis. Future analysis will focus on newly developed bone metabolism markers, as this is a currently evolving area.
* To evaluate body composition in Systemic Lupus Erythematosus utilizing whole body DXA and to determine the contribution of body composition abnormalities to BMD.

Research Design and Method: This study includes a baseline cross-sectional component comparing Systemic Lupus Erythematosus subjects to normal healthy controls followed by a longitudinal follow up study of Systemic Lupus Erythematosus subjects. Systemic Lupus Erythematosus subjects and controls will be evaluated in a single-day visit to the University of California, San Francisco Pediatric Clinical Research Center for clinical assessment and phlebotomy followed by a radiologic evaluation at the Department of Radiology.

ELIGIBILITY:
Inclusion criteria:

* Systemic Lupus Erythematosus subjects 4/11 of the American College of Rheumatology criteria for SLE (23), age less than 22 years.

Exclusion Criteria:

* Neonatal SLE or drug-induced Systemic Lupus Erythematosus
* Subjects who are pregnant, and subjects weighing over 300 pounds, as the densitometry techniques are not reliable above this weight.
* Subjects receiving calcium or vitamin D supplementation will not be excluded but this information will be recorded and evaluated further in the dietary/nutritional assessment.

Ages: 7 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with SLE
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 1999-07-21 (Actual); Primary Completion 2004-07-09 (Actual); Study Completion 2004-07-09 (Actual)

PRIMARY OUTCOMES:
Evaluate whether weak bones are associated with things like medications or amount of fat in muscle | One year
  Bone density measurements by DXA

SECONDARY OUTCOMES:
Evaluate whether weak bones are associated with things like medications or amount of fat in muscle | one year
  Bone density measurements by computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Emily von Scheven, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States